CLINICAL TRIAL: NCT02895919
Title: Is Bedside Inoculation of Ascitic Fluid in Diagnostic Paracentesis Associated With a Higher Sensitivity for Positive Cultures? Prospective Observational Trial
Brief Title: Bedside Inoculation of Ascitic Fluid in Diagnostic Paracentesis
Status: Withdrawn | Type: Observational
Why Stopped: IRB expired
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Other Study IDs: PRO00027101
Record Dates: First submitted 2016-08-31; First posted 2016-09-12 (Estimated); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Ascites; Peritonitis
MeSH Terms: conditions — Ascites; Peritonitis | interventions — Culture Techniques

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Control group - blood culture bottles: Standard of care group for control - will inoculate all samples in blood culture bottles for ascitic fluid culture
  Interventions: Other: Culture
- Study group - sample to lab for culture: Study group - will send a sample of ascitic fluid to lab for inoculation in addition to control sample
  Interventions: Other: Culture

INTERVENTIONS:
Other: Culture — culture of ascitic fluid in standard culture media of blood culture bottles at bedside and fluid collected for culture in laboratory (study arm).

SUMMARY:
This study seeks to determine non inferiority of direct inoculation of ascitic fluid in lab as compared to current culture media standard, bedside inoculation with blood culture bottles.

DETAILED DESCRIPTION:
The purpose of this study is to validate the principal study that recommends inoculation with blood culture bottles at bedside versus lab inoculation (delayed inoculation) of ascitic fluid in the diagnosis of spontaneous bacterial peritonitis. This study had a small sample size (29) and goal is to validate results with a larger sample size. The aim of current proposed study is to assess for non inferiority of lab inoculation of ascitic fluid culture versus current standard of blood culture bottles. To achieve 90% power and true sensitivity 95%, goal is to enroll 460 patients within the course of a year or until number of samples is reached, with plan to compare the sensitivity of bedside inoculation of blood culture bottles versus the lab using sterile plate techniques as per current lab culture technique. Unlike previous study, all comers for ascitic fluid collected will be analyzed that are to undergo diagnostic paracentesis.

ELIGIBILITY:
Inclusion Criteria:

* Ascites on ultrasound

Exclusion Criteria:

* Consent declined

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient population will include all patients undergoing diagnostic paracentesis comparing standard culture protocol (bedside inoculation of blood culture bottles with ascitic fluid) with an additional culture collected for study arm. Patients will be all comers for diagnostic paracentesis.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-08-22 (Actual); Primary Completion 2018-08-19 (Actual); Study Completion 2018-08-19 (Actual)

PRIMARY OUTCOMES:
Growth of bacteria on ascitic fluid culture | through study completion, an average of 1 year to complete enrollment of 460 patients
  Non inferiority of direct inoculation in laboratory as compared to bedside inoculation with blood culture bottles by comparing growth of bacterial growth between both groups, control and study arm.

SECONDARY OUTCOMES:
Time to positive ascitic fluid culture | through study completion, an average of 1 year
  Comparing time to positive culture between control and study arm

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Franco Sadud, MD, Principal Investigator — Medical College of Wisconsin

IPD SHARING:
Plan to Share IPD: Yes